CLINICAL TRIAL: NCT06782802
Title: Clinical Significance and Prognostic Value of Prenatal Diagnosis of Obliteration of the Cavum Septum Pellucidum
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: CSP21
Record Dates: First submitted 2024-12-03; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-10

CONDITIONS: Fetal Neurodevelopmental Disorder; Cavum Septum Pellucidum
Keywords: Cavum septum pellucidum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this observational study is to evaluate the incidence of the occurrence of additional abnormalities in fetuses diagnosed with cavum septum pellucidum (CSP) obliteration performed at second-trimester ultrasound, as well as to analyze the postnatal neurological outcome.

DETAILED DESCRIPTION:
In cases of failure to visualize the CSP (obliterated or absent) and additional brain anatomical abnormalities, the feto-neonatal prognosis turns out to be mainly related to the type of associated malformation. It is still debated, however, the prognosis of an absent or isolated obliteration of the SPC in the presence of remaining regular brain anatomy for the time.

Very often, the patient is offered fetal brain MRI, which, compared with ultrasonography, appears to be endowed with greater accuracy in identifying any additional associated cerebral animals. In our center, it is a shared custom to routinely offer the patient the option of performing an MRI, in all cases of failure to visualize the SPC.

If obliteration of the CSP is confirmed as isolated, normal clinical practice is to perform monthly ultrasound monitoring and a second MRI at approximately 30 to 32 weeks, with the aim of ruling out the appearance of further developmental abnormalities. In addition, a specialized pediatric evaluation is usually performed after birth with the aim of following the child developmentally.

In a retrospective manner, clinical data of patients followed at our center from 01/01/2024 to 31/05/2021, with a finding of obliteration of the CSP at the second trimester, will be considered. Of these patients, data from the morphologic ultrasound and concomitant neurosonography and subsequent MRI (if performed) will be analyzed, as well as those that emerged during follow-ups performed until the end of pregnancy. For the purpose of assessing the fetal neurological outcome, such patients will be contacted by telephone, the study will be explained to them, and a proposal will be made for a psychiatric examination at the department of child neuropsychiatry for their child. During this visit the child will be administered psycho-aptitude tests routinely used, according to normal clinical practice, in neurodevelopmental assessment, in accordance with the child's age.

If the patients do not agree to have their children undergo this visit, only the analysis of the data collected during the visits, performed during pregnancy, will be done.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant participants with a diagnosis of cavum septum pellucidum obliteration made at second-trimester morphologic ultrasound between 19+0 and 21+6 weeks
* Age > or = 18 years at the time of outpatient access
* Acquisition of informed consent form, from the patient and minor
* Patients followed at our center

Exclusion Criteria:

* None

Ages: 28 Days to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants followed at our center between 01/01/2014 and 31/05/2021 with a morphologic ultrasound showing an obliteration of the cavum septum pellucidum will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the incidence of brain abnormalities | During second-trimester ultrasound
  Evaluation of the incidence of associated brain abnormalities, diagnosed by neurosonography and MRI, both at the time of diagnosis and found at subsequent planned follow-ups until the end of pregnancy in fetuses with a finding of obliteration of the cavum septum pellucidum

CONTACTS AND LOCATIONS:
Overall Officials: Gianluigi Pilu, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy